CLINICAL TRIAL: NCT04278079
Title: Evaluation of Pars Plana Vitrectomy With Internal Limiting Membrane Peeling for Myopic Traction Maculopathy
Brief Title: Vitrectomy With Internal Limiting Membrane Peeling for Myopic Traction Maculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sharif Yousef El Emam, Clinical Associate Professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUORU001
Record Dates: First submitted 2020-02-12; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Myopic Traction Maculopathy; Pars Plana Vitrectomy; Internal Limiting Membrane Peeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pars Plana Vitrectomy with Internal Limiting Membrane peel — Pars plana vitrectomy with staining and peeling of internal limiting membrane

SUMMARY:
Investigate the effectiveness and safety of pars plans vitrectomy, with internal limiting membrane peeling for cases of myopic traction maculopathy

DETAILED DESCRIPTION:
Performing pars plana vitrectomy for highly myopic patients with decreased visual acuity is the standard of care for patients with myopic traction. A variety of findings are seen by Optical Coherence Tomography. Epiretinal membranes, retinoschisis, lamellar macular holes, and full thickness macular holes are seen. Undergoing vitrectomy, with or without tamponade, in our center, is retrospectively evaluated. Visual acuity change, as well as improvement of the retinal structure by OCT will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Highly myopic patients, having a refractive errors (spherical equivalent) of more than - 8 Diopter, or an axial length more than 26.5 mm.
* Best Corrected Visual Acuity less than 0.1
* Spectral Domain Optical Coherence Tomography showed; staphylomatous changes, with either: Macular retinoschisis, foveal retinal detachment, full thickness macular hole (with or without macualr hole retinal detachment), or lamellar macular hole, with epiretinal membrane

At least 6 months follow-up

Exclusion Criteria:

* Eyes with diffuse chorioretinal macular atrophy
* Concomitant presence of a choroidal neovascular membrane
* Young patients less than 21 years old.
* History of trauma
* Dense media opacity (corneal/ lenticular)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Improvement of best corrected visual acuity | 6 months

IPD SHARING:
Plan to Share IPD: No